CLINICAL TRIAL: NCT02481453
Title: Étude de l'Effet de la Rapamycine Sur la Force Musculaire et la réponse Immunitaire au Cours de la Myosite à Inclusions: étude RAPAMI"
Brief Title: Rapamycine vs Placebo for the Treatment of Inclusion Body Myositis
Acronym: RAPAMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C12-66; 2013-003485-14 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-06-25 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2017-01

CONDITIONS: Inclusion Body Myositis (IBM)
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapamycin (Experimental): rapamycin 1 mg/ml oral solution, 2 mg/day (2 ml/day), once a day, during one year
  Interventions: Drug: Rapamycin
- Placebo (Placebo Comparator): Placebo oral solution, 2 ml/day, once a day, during one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapamycin — Experimental: rapamycin oral solution, 2 mg/day during one year Comparator: placebo
  Other Names: Sirolimus; Rapamune
  Arms: Rapamycin
Drug: Placebo — Comparator: placebo
  Other Names: Phosal
  Arms: Placebo

SUMMARY:
Sporadic Inclusion Body Myositis (IBM) is the most frequent inflammatory myopathy in patients over 50. It is a slowly progressive, but today untreatable (notably by classical immunosuppressants) disease.

Rapamycin used in organ transplantation blocks the activity of T effector cells, preserves T regulatory cells and induces autophagy (protein degradation), all parameters impaired during IBM.

RAPAMI is a prospective, randomised, controlled, double blind, monocentric, phase IIb trial evaluating rapamycine against placebo.

ELIGIBILITY:
Inclusion Criteria:

* IBM defined by the Benveniste & Hilton-Jones ( Neuromuscul Disord. 2010;20: 414-21) or Llyod criteria (Neurology 2014; 83: 426-433)

Exclusion Criteria:

* Impossiblility to walk 10 meters
* Hypersensitivity to rapamycin or one compound of the oral solution
* Severe respiratory insufficiency (FVC < 50% and/or FEV1 < 50%)
* Severe chronic kidney disease (Estimated Glomerular Filtration Rate < 15 ml/min and/or proteinuria > 0.3 g/24h)
* Chronic liver disease (cirrhosis and/or ALT/AST > 2.5 normal values)
* Cancer non in remission (necessitating specific treatment) during the past 12 months
* Connective Tissue Disease non in remission (necessitating specific treatment) during the past 12 months
* Pregnancy
* Seropositivity for HIV, HCV or HBV
* Total cholesterolemia > 8 mmol/l
* Triglyceridemia > 5 mmol/l
* Hemoglobinemia < 11 g/dL
* Thrombopenia < 100 000/mm3
* Neutropenia < 1500/ mm3
* Lymphopenia < 1000/ mm3

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
stabilization of quadiceps strength measured by myometry | 52 weeks

SECONDARY OUTCOMES:
stabilization of hand grip strength measured by myometry | 52 weeks
comparison of 6 minutes walking test | 52 weeks
composite measure of the handicap | 52 weeks
  Rivermead Mobility Index (RMI), scale Walton, Inclusion Body Myositis Weakness Composite Index (IBMWCI), Inclusion Body Myositis Functional rating scale (IBMFRS)
Quality of life by different scales | 52 weeks
  Health Assessment Questionnaire (HAQ), Instrumental activities of daily living (IADL),Individualized Neuromuscular Quality of Life Questionnaire (INQol)
measures of muscle fatty replacement by MRI | 52 weeks
Measure of the tolerance | 52 weeks
  Efficacy will be measured by:
  check list of the known side effect of rapamycin.
measure of inflammation by MRI | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Paris Est _Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benveniste O, Hogrel JY, Belin L, Annoussamy M, Bachasson D, Rigolet A, Laforet P, Dzangue-Tchoupou G, Salem JE, Nguyen LS, Stojkovic T, Zahr N, Hervier B, Landon-Cardinal O, Behin A, Guilloux E, Reyngoudt H, Amelin D, Uruha A, Mariampillai K, Marty B, Eymard B, Hulot JS, Greenberg SA, Carlier PG, Allenbach Y. Sirolimus for treatment of patients with inclusion body myositis: a randomised, double-blind, placebo-controlled, proof-of-concept, phase 2b trial. Lancet Rheumatol. 2021 Jan;3(1):e40-e48. doi: 10.1016/S2665-9913(20)30280-0. Epub 2020 Oct 12. PMID 38273639
- [Background] Benveniste O, Hilton-Jones D. International Workshop on Inclusion Body Myositis held at the Institute of Myology, Paris, on 29 May 2009. Neuromuscul Disord. 2010 Jun;20(6):414-21. doi: 10.1016/j.nmd.2010.03.014. Epub 2010 Apr 21. No abstract available. PMID 20413309
- [Background] Lloyd TE, Mammen AL, Amato AA, Weiss MD, Needham M, Greenberg SA. Evaluation and construction of diagnostic criteria for inclusion body myositis. Neurology. 2014 Jul 29;83(5):426-33. doi: 10.1212/WNL.0000000000000642. Epub 2014 Jun 27. PMID 24975859